CLINICAL TRIAL: NCT05234697
Title: Effect of Daytime Variation on Postoperative Hyperalgesia Induced by Opioids
Status: Completed | Type: Observational
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Postoperative hyperalgesia
Record Dates: First submitted 2022-01-12; First posted 2022-02-10 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Postoperative Hyperalgesia
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood is collected before and after the surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Morning group: Surgery performed during 08:00 to 12:00
  Interventions: Drug: Remifentanil
- Afternoon group: Surgery performed during 14:00 to 18:00
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — Remifentanil was used for maintenance of anesthesia.

SUMMARY:
To explore the effect of daytime variation on postoperative hyperalgesia induced by opioids. Patients receiving endoscopy surgery under general anesthesia during 08:00-12:00(morning group, n=30) and 14:00-18:00(afternoon group, n=30) using remifentanil for anesthesia maintenance were respectively included. Postoperative hyperalgesia at PACU and 24 hours after surgery were assessed through mechanical pain measurement. Comparative analysis of postoperative hyperalgesia levels, pain and analgesic requirements between morning group and afternoon group were performed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classification I-II
* Abdominal endoscopy surgery
* Estimated surgery duration 1-2h
* Right handedness
* Voluntarily receive postoperative intravenous controlled analgesia

Exclusion Criteria:

* Heavy smoking or alcohol dependence
* Puerpera or lactation women
* History of chronic pain
* Analgesic use within one month before surgery
* Allergy to opioids
* Can not follow with the study procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving endoscopy surgery under general anesthesia during 08:00-12:00(morning group, n=30) and 14:00-18:00(afternoon group, n=30) using remifentanil for anesthesia maintenance were included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Postoperative hyperalgesia when discharged from postanesthesia care unit | from the 30 minutes before the surgery until to the time when discharged from postanesthesia care unit, assessed up to about 2 hours
  The ratio of pressure pain threshold when discharged from PACU compare to before surgery

SECONDARY OUTCOMES:
Postoperative hyperalgesia at 24 hours after surgery | from the 30 minutes before the surgery until to 24 hours after surgery
  The ratio of pressure pain threshold at 24 hours after surgery compare to before surgery
Postoperative pain intensity | from the time when the surgery was completed until to 24 hours after surgery
  Pain intensity was assessed by numerical rating scale (0-10, 0 represents painless; 10 represents intolerable pain)
Postoperative analgesic requirements | from the time when the surgery was completed until to 24 hours after surgery
  Analgesic requirements was assessed by recording the volume of patient controlled analgesia pump
Plasma concentration of remifentanil and sufentanil | from 30 minutes before the surgery until to the time after stop infusion of remifentanil, assessed up to about 2 hours
  Determined by Elisa test
Activity of plasma nonspecific esterase | from 30 minutes before the surgery until to the time after stop infusion of remifentanil, , assessed up to about 2 hours
  Determined by laboratory detection

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, The Second Affiliated Hospital, Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data for this study is available from the sponsor on reasonable request through email.

REFERENCES:
- [Derived] Shu B, Liu H, Zheng X, He J, Wu Y, Chen J, Chen Y, Tian H, Ju D, Huang H, Duan G. Opioid infusions at different times of the day produce varying degrees of opioid-induced hyperalgesia. Br J Anaesth. 2023 Dec;131(6):1072-1081. doi: 10.1016/j.bja.2023.08.039. Epub 2023 Oct 9. PMID 37821342